CLINICAL TRIAL: NCT01813084
Title: A Randomised, Double Blind, Placebo-controlled, Three Part Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Treatment With Single and Repeat Doses of Inhaled RV1729 in Healthy Subjects and Subjects With Mild to Moderate Asthma
Brief Title: A Study to Investigate the Safety, Tolerability and Pharmacokinetics of Single and Repeat Doses of RV1729
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Respivert Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STN001; 2012-005452-42 (EudraCT Number)
Record Dates: First submitted 2013-03-14; First posted 2013-03-18 (Estimated); Last update posted 2014-04-24 (Estimated); Status verified 2014-04

CONDITIONS: Asthma; Healthy Volunteers
MeSH Terms: conditions — Asthma | interventions — 6-(2-((4-amino-3-(3-hydroxyphenyl)-1H-pyrazolo(3,4-d)pyrimidin-1-yl)methyl)-3-(2-chlorobenzyl)-4-oxo-3,4-dihydroquinazolin-5-yl)-N,N-bis(2-methoxyethyl)hex-5-ynamide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Part A: single dose escalation (Experimental)
  Interventions: Drug: RV1729 single dose; Drug: RV1729 matching placebo single dose
- Part B: 14 day repeat dose escalation (healthy volunteers) (Experimental)
  Interventions: Drug: RV1729: 14 day repeat dose; Drug: RV1729 matching placebo: 14 day repeat dose
- Part C: 14 day repeat dose (asthma patients) (Experimental)
  Interventions: Drug: RV1729: 14 day repeat dose; Drug: RV1729 matching placebo: 14 day repeat dose

INTERVENTIONS:
Drug: RV1729 single dose — Safety and tolerability of single escalating doses
  Arms: Part A: single dose escalation
Drug: RV1729 matching placebo single dose — Safety and tolerability of single escalating doses
  Arms: Part A: single dose escalation
Drug: RV1729: 14 day repeat dose — Safety and tolerability of repeat escalating doses
  Arms: Part B: 14 day repeat dose escalation (healthy volunteers); Part C: 14 day repeat dose (asthma patients)
Drug: RV1729 matching placebo: 14 day repeat dose — Safety and tolerability of repeat escalating doses
  Arms: Part B: 14 day repeat dose escalation (healthy volunteers); Part C: 14 day repeat dose (asthma patients)

SUMMARY:
RV1729 is a new medicine being developed for possible treatment of asthma and smoking related lung disease (also known as chronic obstructive pulmonary disease - COPD).

The main purpose of this study is to investigate the safety, tolerability and pharmacokinetics of single and repeat doses of RV1729.

ELIGIBILITY:
Inclusion Criteria:

* Be a man or woman between 18 to 50 years of age, inclusive, at the time of signing the informed consent
* Sign an informed consent document indicating they understand the purpose of and procedures required for the study and are willing to participate in the study
* If a woman of childbearing potential, must have a documented menstrual period prior to the first dose and be willing and able to use two forms of contraception from screening to 90 days after the final dose of RV1729, OR
* If a woman of non-childbearing potential must be amenorrhoeic for greater than 1 year or have been permanently sterilised, OR
* If a man, must be willing and able to use one of the contraception methods listed in the protocol and agree not to donate sperm, the first dose until 90 days after they receive the final dose of RV1729.
* Body mass index between 19 and 30 kg/m2 (inclusive), and body weight not less than 50 kg
* Vital sign assessments within normal ranges: blood pressure between 90 and 140 mmHg systolic, inclusive, and between 40 and 90 mmHg diastolic; heart rate 40 - 100 bpm
* Have a 12-lead ECG consistent with normal cardiac conduction and function
* Capable of complying with all study restrictions and procedures including ability to use the study Dry Powder Inhaler correctly

Parts A & B (healthy volunteers only)

* Healthy as determined by a physician, based on a full medical evaluation including medical history, physical examination, laboratory tests.
* Prebronchodilator spirometry readings (FEV1 and FVC) to be ≥ 80% predicted value and FEV1/FVC ratio > 0.7 at screening
* Are not taking prescription medications for 14 days prior to screening and agree not to use prescription medications throughout the duration of the study.
* Not taking over the counter medications for 14 days prior to Screening visit to the final follow up visit

Part C (asthma patients only)

* Documented history of asthma, for at least 6 months prior and currently being treated with as needed short-acting beta -agonist therapy and daily inhaled corticosteroids
* Have a diagnosis of asthma. This may be confirmed with bronchodilator reversibility or a challenge test.
* Have a pre-bronchodilator forced expiratory volume in the first second (FEV1) ≥ 65% of predicted normal value
* Treated with a stable low or medium dose of inhaled corticosteroid for at least 4 weeks prior to screening
* Have stable asthma based on physician assessment at screening with no asthma exacerbation requiring augmentation of therapy in the 12 weeks prior to screening and no hospitalisation for asthma in the 5 years prior to screening
* Not have a clinical abnormality or laboratory parameters outside the reference range for the population being studied
* Not taking over the counter (OTC) medications and herbal medication for 14 days prior to screening visit and up to the final follow up visit

Exclusion Criteria:

* Upper or lower respiratory tract infection within 4 weeks of the screening visit
* Clinically significant abnormal values for haematology, clinical chemistry or urinalysis at screening
* History of, or a reason to believe a subject has a history of drug or alcohol abuse within the past 5 years
* Positive test for alcohol or drugs of abuse at screening or prior to dosing
* History of clinically significant allergies that would contraindicate participation
* Known allergy to the study drug or any of the excipients of the formulation
* Donated blood or blood products or had substantial loss of blood (more than 500 mL) within 3 months before the study
* Received an experimental drug or used an experimental medical device within 3 months or within a period less than 10 times the drug's half life before the first dose of the study drug is scheduled
* If a woman, has a positive serum pregnancy test at screening or on admission, is pregnant, breast-feeding or planning to become pregnant during the study
* Positive test for human immunodeficiency virus (HIV) 1 and 2 antibodies, hepatitis B virus (HBV) infection, or hepatitis C antibodies
* History of smoking or use of nicotine-containing substances within the previous 6 months, or a positive carbon monoxide test at screening
* Preplanned surgery or procedures that would interfere with the conduct of the study
* Employee of the investigator or study center, with direct involvement in the proposed study or other studies under the direction of that investigator or study center, as well as family members of the employees or the investigator.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities
* History of regular alcohol consumption within 6 months of the study
* The subject is unable or unwilling to comply fully with the study protocol
* Subject is mentally or legally incapacitated
* Unable or unwilling to undergo multiple venepuncture procedures or the subject has poor access to veins suitable for cannulation
* Any other reason that the Investigator considers makes the subject unsuitable to participate

Part C (asthma patients only)

* Administration of oral, injectable or dermal steroids within 3 months or intranasal steroids within 1 week of the screening visit.
* Has ever had an episode of life-threatening asthma
* Any acute or chronic illness or clinically relevant abnormality other than asthma
* Use of Cysteine within 24 hours of screening and throughout the study period
* Has severe asthma based on Investigator assessment

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2013-05; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment emergent adverse events | Cohort 1, 49 days: Cohorts 2 & 3, 21 days; Cohorts 4, 5, 6 & 7, 28 days
  Assessment of the number of adverse events reported by subjects following dosing.
ECG Assessment (12-lead ECG) | Cohort 1, 49 days: Cohorts 2 & 3, 21 days; Cohorts 4, 5, 6 & 7, 28 days
  Change from pre-dose values.
Vital sign assessment (blood pressure & heart rate) | Cohort 1, 49 days: Cohorts 2 & 3, 21 days; Cohorts 4, 5, 6 & 7, 28 days
  Change from pre-dose values.
Spirometry assessment (FEV1 & FVC) | Cohort 1, 49 days: Cohorts 2 & 3, 21 days; Cohorts 4, 5, 6 & 7, 28 days
  Change from pre-dose values
Clinical laboratory assessments (blood and urine samples) | Cohort 1, 49 days: Cohorts 2 & 3, 21 days; Cohorts 4, 5, 6 & 7, 28 days
  Change from pre-dose values

SECONDARY OUTCOMES:
Plasma RV1729 levels | Cohort 1: Day 1 (0,10,15&30min,1,2,4,6&24h), 5 treatment periods. Cohorts 2&3: Day 1 (0,10,15&30min 1,2,4,6,8,12h), Days 2-8 (24,48,72,96,120,144&168h). Cohorts 4,5,6&7: Days 1, 7&14 (0,10,15&30min,1,2,4,6,8,10,12&24h) & Days 8-13 & 16-21 & 28 (0h)

OTHER OUTCOMES:
Serum biomarkers (measuring markers of inflammation in the blood) | Cohorts 4, 5, 6 & 7: Days 1 & 14 (0, 4 & 24 h), Day 4 (0 h) and Day 28
Exhaled Nitric Oxide (measuring airway inflammation) | Cohorts 4, 5, 6 & 7: Screening then Days 1 & 4 (0 h), Day 14 (0, 1 & 24 h)
Exhaled breath condensate (measuring markers of oxidative stress) | Cohorts 4, 5, 6 & 7: Screening then Days 1 & 14 (0 & 6 h)
Urinary cortisol, 4-beta hydroxycholesterol and Leukotriene E4 (LTE4) | Cohorts 4, 5, 6 & 7: Days -1 & 14 (0 to 24 h collection)
Sputum cells and biomarkers (measuring markers of inflammation in found in sputum) | Cohorts 6 & 7: Screening then Day 14 (6 h)

CONTACTS AND LOCATIONS:
Overall Officials: Jerome Boscia, MD, Study Director — Sponsor GmbH
Locations (2):
- United Kingdom (2):
  - London
  - Manchester